CLINICAL TRIAL: NCT06702267
Title: 23001, Clinical Precision and In-use Analyte Stability Study for Four (4) Parameters in Neonate Arterial Blood for PICO70 and SafePICO
Brief Title: Clinical Precision and In-use Analyte Stability Study for Four (4) Parameters in Neonate Arterial Blood for PICO70 and SafePICO
Status: Completed | Type: Observational
Sponsor: Radiometer Medical ApS (Industry)
Responsible Party: Sponsor
Other Study IDs: DC-086959
Record Dates: First submitted 2024-07-09; First posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Measure the Precision and Stability in PICO70 and SafePICO Over Time

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples collected from cord/placenta and destroyed immediately after measurements.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- cord/placenta from women given birth: One single group is included in the study for the investigation of the PICO70 and safePICO syringes.
  Interventions: Device: arterial blood samplers with needles PICO70 and safePICO syringes.

INTERVENTIONS:
Device: arterial blood samplers with needles PICO70 and safePICO syringes. — PICO70 is a self-filling syringe for sample volumes in the range of 0.3-1.5 mL. All syringes are delivered with needle cube for safe needle disposal and a standard tip cap to reduce the risk of blood contact during blood mixing and sample transportation.
  safePICO is a more advanced group of syringes based on the PICO70 family. They contain a gold coated magnetic steel ball facilitating automatic mixing of the blood when being used with the Radiometer ABL 90 with mixing module. The safePICO is a self-filling syringe covering a volume range of 0.7-1.5 mL and includes a vented safe tip cap (VTC), which simplifies removal of air bubbles and avoid the operator to get in contact with the blood, after attachment to the syringe. Some variants of safePICO are delivered with a needle shield device (NSD) to ensure safe removal of the needle.

SUMMARY:
The objective is to determine the total (within-lot and between lots) precision for four (4) parameters (pO2, tBil, ctHb and FHbF) in neonatal arterial blood. Furthermore, the objective is to determine the analyte in-use stability for each blood gas syringe in arterial blood for neonatal blood parameters.

In-use analyte stability in neonatal arterial blood in PICO70 and safePICO for each parameter, measuring at four testing timepoints.

It is expected that he precision performance of each parameter is equal to or within the acceptance criteria/performance claim.

The in-use analyte stability measured at four testing timepoint is within the acceptance criteria.

DETAILED DESCRIPTION:
The study is a Post-Market Clinical Follow-up (PMCF) randomized unblinded study, to be conducted across two sites in Denmark, using subject whole blood samples from Umbilical cord/placenta to determine the precision and stability for the PICO70/safePICO syringes when measuring four parameters using the RMED ABL90 FLEX PLUS analyzer.

For PICO70 + safePICO: 40 + 40 completed arterial series of samples consisting of 5 syringes are needed: The syringes will be from three different lots (A,B,C) and analyzed at four different time points, T0 min., T15 min., T30 min., T45 min. to cover measurements completed within 0 - 45 minutes.

Both PICO70 and safePICO arterial blood series of samples can be drawn from one subject/placenta, which brings a range of 40 - 80 completed subjects enrolled in total for the study. If subjects are enrolled but not completed according to the protocol such subject will need replacement. Whole blood will be collected from subject cord/placenta in a mother syringe and distributed when relevant into the five (5) PICO70 and five (5) safePICO syringes for measurments.

It can be relevant to collect venous blood if sufficient volume of arterial blood is not available for the cord/placenta blood collection.

The mother syringe will be heparinized. The amount of heparin in the mother syringe will be determined based on the total volume of the samples.

Series of syringes will be randomized and provided to site in kits of 5 marked syringes prior to study start to get an unbiased precision result. Three different Lot numbers for both the PICO70 and safePICO syringes are to be analyzed during the conduct of the study. The order of the three Lots (ABC) to be analyzed are randomized and included in each Kit. Each kit will be marked with subject number and randomization number. Site has to use each kit for the next subject in subject number order (101, 102, 103 etc.). The 5 syringes will each be marked as follow; 1T0, 2T0, 3T15, 4T30 and 5T45 which indicates when and in what order the samples shall be measured after samples are drawn and contrived for specific level. T0 shall be measured within 10 min. after contriving is completed.

The four (4) parameters pO2, tBil, ctHb and FHbF will be analysed for each syringe in the syringe series. Three parameters (pO2, tBil, FHbF) will be contrived according to guideline. The contriving procedure will be performed either by the site or lab technician. The contriving of the two parameters pO2 and tBil will be measured together with ctHb. FHbF will be analyzed in a separate sample after being contrived.

ELIGIBILITY:
Inclusion Criteria:

Subject must be 18 years of age or older Subject must be pregnant and at least 37 weeks of gestation Subject must be admitted to the hospital maternity ward to give birth vaginally or to undergo cesarian section. Subject must be evaluated by the principal investigator or designee as suitable for the study according to the protocol

Exclusion Criteria:

Subjects already enrolled in the study Subjects exposed to either Fluorescein dye or Patent Blue dye with last dose within 72 hours, should be excluded due to potential interference.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Subject must be pregnant and at least 37 weeks of gestation.
Study Population: Pregnant adult women 18 years of age or older admitted to the maternity ward to give birth vaginally or to undergo cesarian section after 37 weeks of gestation. The pregnant woman gives informed consent to ensure accept of the cord/placenta sample collection and handling procedures. No study related procedures will be completed for the pregnant woman.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2023-12-12 (Actual); Primary Completion 2024-03-04 (Actual); Study Completion 2024-03-04 (Actual)

PRIMARY OUTCOMES:
In-use analyte stability in neonatal arterial blood in PICO70 and safePICO for each parameter, measuring at four testing timepoints. | One subject delivers blood samples to be measured over time (45 min.)
  Furthermore, the objective is to determine the analyte in-use stability for each blood gas syringe in arterial blood for neonatal blood parameters.
Precision in neonatal arterial blood in PICO70 and safePICO for each parameter. | One subject delivers blood samples to be measured over time (45 min.)
  The objective is to determine the total (within-lot and between lots) precision for four (4) parameters (pO2, tBil, ctHb and FHbF) in neonatal arterial blood.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Jeppegaard, PI, Principal Investigator — External Coordinating Principal Investigator
Locations (1):
- Hvidovre Hospital, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: Yes
The study results will be available to participating Investigators and to support The results are also available for supporting the safety and performance of the arterial blood syringes with needles, PICO70, safePICO70 and safePICO self-fill according to requirements.
Supporting Information: CSR
Time Frame: 4 months in Q4 2023 - Q1 2024. Data will become available in Feb./March 2025